CLINICAL TRIAL: NCT05436275
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of CM310 in Patients With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: A Study of CM310 in Patients With Chronic Rhinosinusitis With Nasal Polyposis （CROWNS-2）
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-102208
Record Dates: First submitted 2022-06-20; First posted 2022-06-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyposis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 (Experimental): CM310 300mg is given subcutaneously (SC) every two weeks
  Interventions: Biological: Placebo
- Placebo (Placebo Comparator): Placebo is given subcutaneously (SC) every two weeks
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — 300 mg every two weeks
  Arms: Placebo
Biological: Placebo — once every two weeks
  Arms: CM310

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled Phase III study to evaluate the efficacy and safety of CM310, and to observe the life quality of subjects, the Pharmacokinetics, Pharmacodynamics and immumogenicity of CM310 in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP).

DETAILED DESCRIPTION:
The study consists of a Screening Period (up to 4 weeks), Treatment Period (24 weeks for double-blind treatment period and 28 weeks for open-label maintenance treatment) and Safety Follow-up Period (8 weeks).

180 patients who meet eligibility criteria will be randomized 1:1 to receive either CM310 300 mg or matched placebo subcutaneously every two weeks (Q2W) for a total of 12 times at the double-blind treatment period and 14 times at the open-label treatment period. All patients will receive MFNS on a daily basis as a background treatment throughout the study.

Central reading will be implemented to nasal endoscopic nasal polyp score (NPS) , CT scans to Lund-Mackay score and volume of the involved area of nasosinusitis on 3D-construction images, and nasal polyp biopsy tissue analysis to eosinophil counts & percentage.

ELIGIBILITY:
Inclusion Criteria:

* with chronic rhinosinusitis with nasal polyposis (CRSwNP).
* Nasal Polyp Score (NPS) of ≥5 with a minimum score of 2 in each nasal cavity.
* NCS score of 2 or 3 at screening period, and at least 2 at baseline.
* Contraception.

Exclusion Criteria:

* Not enough washingout period for previous therapy, e.g., less than 10 weeks or 5 half-lives (whichever is longer) for IL-4Rα antagonists, less than 8 weeks or 5 half-lives for biologic therapy/systemic immunosuppressant, less than 6 months for sinus surgery (including polypectomy).
* Participated and any studies of CM310.
* With malignant or benign tumor of nasal cavity.
* Vaccination with live attenuated vaccine within 12 weeks before randomization or during the planned study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Nasal Polyps Score (NPS) | at week 24
  Change from baseline in the Nasal Polyps Score (NPS) at week 24. NPS score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Nasal Congestion Score (NCS) | at week 24
  Change from baseline in the Nasal Congestion Score (NCS) at week 24. NCS score range from 0 to 3, with higher score means worse nasal symptom.

SECONDARY OUTCOMES:
Safety parameters | Baseline up to Week 60
  Incidence of treatment-emergent adverse events (TEAEs).
Pharmacokinetics (PK) | Baseline up to Week 60
  Concentration of CM310 in serum
Pharmacodynamics (PD) | Baseline up to Week 60
  Change from baseline in serum biomarker level (Thymus- and activation-regulated chemokine).
Anti-drug antibodies (ADA) | Baseline up to Week 60
  Incidence of ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shen S, Yan B, Wang M, Wu D, Piao Y, Tang J, Yang X, Cao Z, Xue J, Liu W, Liu S, Shi L, Wang G, Song X, Lu Y, Chen J, Jiang L, Ye J, Yu S, Yang Y, Fang H, Li J, Shi H, Fan J, Yan H, Wang H, Chen B, Wang C, Zhang L; CROWNS-2 Study Investigators. Stapokibart for Severe Uncontrolled Chronic Rhinosinusitis With Nasal Polyps: The CROWNS-2 Randomized Clinical Trial. JAMA. 2025 Aug 18;334(11):962-72. doi: 10.1001/jama.2025.12515. Online ahead of print. PMID 40824573
- [Derived] Shen S, Yan B, Wang M, Wu D, Wang C, Zhang L. Anti-IL-4Ralpha monoclonal antibody (CM310) in patients with chronic rhinosinusitis with nasal polyps (CROWNS-2): Rationale and design of a multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Asia Pac Allergy. 2024 Aug;14(3):118-123. doi: 10.5415/apallergy.0000000000000156. Epub 2024 Aug 5. PMID 39220573